CLINICAL TRIAL: NCT05698420
Title: Investigation of the Effects of Medium Cut-off Dialyzers Versus High-Flux Dialyzers on Clinical and Laboratory Parameters of Prevalent Hemodialysis Patients
Status: Completed | Type: Observational
Sponsor: Sanliurfa Mehmet Akif Inan Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Tuncay Sahutoglu, Associate Professor, Sanliurfa Mehmet Akif Inan Education and Research Hospital
Other Study IDs: MCOx_MAIEAH_001
Record Dates: First submitted 2023-01-05; First posted 2023-01-26 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Hemodialysis-Associated Pruritus; Malnutrition-Inflammation-Cachexia Syndrome; Restless Legs Syndrome; Anemia of Chronic Kidney Disease; Depressive Disorder
MeSH Terms: conditions — Restless Legs Syndrome; Depressive Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and plasma extracts from venous blood samples were stored at -80C of the hospital.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The Theranova 400 group, also known as the MCO group.: Patients undergoing maintenance hemodialysis will receive dialysis treatment using the Theranova 400 device.
  Interventions: Device: Dialysis using the Theranova-400 device.
- The FX80 group, also known as the high-flux group.: Patients undergoing maintenance hemodialysis will receive dialysis treatment using the FX80 device.
  Interventions: Device: Dialysis using the FX80 device.

INTERVENTIONS:
Device: Dialysis using the Theranova-400 device. — Patients receive hemodialysis treatment using the Theranova-400 dialyzer.
  Groups: The Theranova 400 group, also known as the MCO group.
Device: Dialysis using the FX80 device. — Patients receive hemodialysis treatment using the FX80 dialyzer.
  Groups: The FX80 group, also known as the high-flux group.

SUMMARY:
In this study, the investigators aimed to observe the effects of medium cut-off dialysis filters and high-flux dialysis filters on malnutrition inflammation score, uremic itching, restless leg syndrome, anemia, and ESA treatment, which are prominent complications in hemodialysis, and routine follow-up parameters.

DETAILED DESCRIPTION:
The study is designed as a single-center, prospective, observational research. A total of 50 stable-course chronic hemodialysis patients over 18 years of age and treated for at least 3 months will be included in the study and the study period will be planned for 12 months. 25 of the 50 chronic hemodialysis patients planned to be included in the study will use MCO-membrane and the other 25 will use high-flux membrane. The distribution of patients to the high-flux membrane and MCO membrane groups will be done randomly (sequentially single-pair number method). Then, the standard 12-hour (3x4 hours/week) hemodialysis treatment will continue. At the beginning of the study (0.), at the end of the third (3.) month and at the end of the sixth (6.) month;

Monthly laboratory tests routinely performed on hemodialysis patients (tests routinely performed in hemodialysis patient follow-up) 5 ml blood samples will be taken from the hemodialysis set to determine the levels of medium-large molecule-weight toxins-wastes and inflammatory parameters before and after dialysis, and the sera will be separated and stored at -80oC for use at the end of the study.

Automatic blood pressure measurement will be performed before and after hemodialysis to evaluate arterial stiffness.

The Malnutrition Inflammation Score will be applied to evaluate the nutritional status (the MIS form is given in the appendix) Visual Analog Scale will be used for appetite Visual Analog Scale will be used for uremic pruritus Depression scale screening (Beck's scale)

ELIGIBILITY:
Inclusion Criteria:

* Chronic hemodialysis patients
* Patients continuing the hemodialysis program for at least 3 months
* Patients over 18 years of age

Exclusion Criteria:

* Patients with advanced heart failure, malignancy, terminal illness
* Patients with active infectious disease
* Acute hemodialysis patients
* Patients vascular access dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prevalent patients who are receiving hemodialysis treatment three times a week and are otherwise in stable condition.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Malnutrition-inflammation score (MIS) | Prior to randomization, at the start of the study.
  At the start of the study, the malnutrition-inflammation score will be recorded. This score ranges from 0 to 30, with higher scores indicating worse outcomes.
Malnutrition-inflammation score (MIS) | At the end of the 6th month after randomization.
  The malnutrition-inflammation score will be recorded at the conclusion of the study. This score ranges from 0 to 30, with higher scores indicating worse outcomes.
Depressive disorder | Prior to randomization, at the start of the study.
  At the start of the study, the Beck's depression scale will be recorded. This score ranges from 0 to 63, with higher scores indicating worse depression.
Depressive disorder | At the end of the 6th month after randomization.
  At the conclusion of the study, the Beck's depression scale will be recorded. This score ranges from 0 to 63, with higher scores indicating worse depression.
Uremic pruritus | Prior to randomization, at the start of the study.
  At the start of the study, the visual analog scale for pruritus will be recorded. This score ranges from 0 to 10, with higher scores indicating worse itching.
Uremic pruritus | At the end of the 6th month after randomization.
  At the conclusion of the study, the visual analog scale for pruritus will be recorded. This score ranges from 0 to 10, with higher scores indicating worse itching.
Restless leg syndrome | Prior to randomization, at the start of the study.
  At the start of the study, the Restless Leg Syndrome screening questionnaire will be administered. This score ranges from 0 to 40, with higher scores indicating worse symptoms.
Restless leg syndrome | At the end of the 6th month after randomization.
  At the conclusion of the study, the Restless Leg Syndrome screening questionnaire will be administered. This score ranges from 0 to 40, with higher scores indicating worse symptoms.
Appetite | Prior to randomization, at the start of the study.
  At the start of the study, the visual analog scale of appetite will be recorded. This score ranges from 0 to 5, with higher scores indicating better appetite.
Appetite | At the end of the 6th month after randomization.
  At the conclusion of the study, the visual analog scale of appetite will be recorded. This score ranges from 0 to 5, with higher scores indicating better appetite.
Hemoglobin | March 2020
  Hemoglobin levels will be measured on a monthly basis.
Hemoglobin | April 2020
  Hemoglobin levels will be measured on a monthly basis.
Hemoglobin | May 2020
  Hemoglobin levels will be measured on a monthly basis.
Hemoglobin | June 2020
  Hemoglobin levels will be measured on a monthly basis.
Hemoglobin | July 2020
  Hemoglobin levels will be measured on a monthly basis.
Hemoglobin | August 2020
  Hemoglobin levels will be measured on a monthly basis.
Hemoglobin | September 2020
  Hemoglobin levels will be measured on a monthly basis.
Erythropoietin Doses | March 2020
  Weight-adjusted doses of erythropoietin will be prescribed on a monthly basis.
Erythropoietin Doses | April 2020
  Weight-adjusted doses of erythropoietin will be prescribed on a monthly basis.
Erythropoietin Doses | May 2020
  Weight-adjusted doses of erythropoietin will be prescribed on a monthly basis.
Erythropoietin Doses | June 2020
  Weight-adjusted doses of erythropoietin will be prescribed on a monthly basis.
Erythropoietin Doses | July 2020
  Weight-adjusted doses of erythropoietin will be prescribed on a monthly basis.
Erythropoietin Doses | August 2020
  Weight-adjusted doses of erythropoietin will be prescribed on a monthly basis.
Erythropoietin Doses | September 2020
  Weight-adjusted doses of erythropoietin will be prescribed on a monthly basis.
Phosphorus levels control | March 2020
  Serum phosphorus levels will be tested on a monthly basis.
Phosphorus levels control | April 2020
  Serum phosphorus levels will be tested on a monthly basis.
Phosphorus levels control | May 2020
  Serum phosphorus levels will be tested on a monthly basis.
Phosphorus levels control | June 2020
  Serum phosphorus levels will be tested on a monthly basis.
Phosphorus levels control | July 2020
  Serum phosphorus levels will be tested on a monthly basis.
Phosphorus levels control | August 2020
  Serum phosphorus levels will be tested on a monthly basis.
Phosphorus levels control | September 2020
  Serum phosphorus levels will be tested on a monthly basis.
Parathyroid hormone levels control | March 2020
  Serum parathyroid hormone levels will be tested on a monthly basis.
Parathyroid hormone levels control | April 2020
  Serum parathyroid hormone levels will be tested on a monthly basis.
Parathyroid hormone levels control | May 2020
  Serum parathyroid hormone levels will be tested on a monthly basis.
Parathyroid hormone levels control | June 2020
  Serum parathyroid hormone levels will be tested on a monthly basis.
Parathyroid hormone levels control | July 2020
  Serum parathyroid hormone levels will be tested on a monthly basis.
Parathyroid hormone levels control | August 2020
  Serum parathyroid hormone levels will be tested on a monthly basis.
Parathyroid hormone levels control | September 2020
  Serum parathyroid hormone levels will be tested on a monthly basis.

CONTACTS AND LOCATIONS:
Overall Officials: Tuncay Sahutoglu, M.D., Principal Investigator — Mehmet Akif Inan Training and Research Hospital
Locations (1):
- Mehmet Akif Inan Training and Research Hospital, Sanliurfa, Karaköprü, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No